CLINICAL TRIAL: NCT02779465
Title: Study of Oral Vitamin D Treatment for the Prevention of Hepatocellular Carcinoma in Patients With Chronic Hepatitis B
Brief Title: Oral Vitamin D Treatment for the Prevention of Hepatocellular Carcinoma
Acronym: VDHCC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yutian Chong, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-CYT-VD5010
Record Dates: First submitted 2016-05-13; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis B; Carcinoma, Hepatocellular
Keywords: vitamin D treatment; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular; Hepatitis B, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Drug: Vitamin D3 800 IU daily besides the anti-virus treatment with nucleos(t)ide medicine
  Interventions: Drug: Vitamin D3
- Control (No Intervention): chronic hepatitis B patients with long term anti-virus therapy

INTERVENTIONS:
Drug: Vitamin D3 — Participants with chronic hepatitis B will take 800 IU of vitamin D3 per day by mouth besides the anti-virus treatment with nucleos(t)ide medicine
  Arms: Vitamin D

SUMMARY:
The purpose of this study is to determine whether vitamin D is effective in the prevention of hepatocellular carcinoma in those patients with chronic hepatitis B.

DETAILED DESCRIPTION:
Potential participants will be identified from the follow-up cohort of chronic hepatitis B in the third Affiliated Hospital of Sun Yat-sen University (3rd SYSU). The hepatologists at the 3rd SYSU's Infectious Disease Institute will ask each potential participant if she/he is interested in participating. If the patient expresses an interest in the study, one of the researchers will meet with the patient when he/she is at the 3rd SYSU for a regular appointment and will describe the study to the potential participant. If a patient continues to be interested in participating, she/he will be given a copy of the review board approved consent document to read. The consent document will be used as a guide for explaining the study in detail to the patient. The participant allocated to the experimental group will be contacted by one of the investigators on the research team and instructed to begin taking 2 tablets per day (800 IU total) of vitamin D3 besides their regular anti-virus treatment. Those patients allocated in the control group will be informed that they are not to take any vitamin D3 and they will be followed as controls for this study. The researcher will investigate general treatment benefits and the potential to reduce the development of Hepatocellular carcinoma (HCC), also known as liver cancer. Improvement of treatment benefits will be determined by interviews with patients, the level of HBsAg and HBeAg, the development of liver fibrosis and evidence of HCC on routine imaging.

ELIGIBILITY:
Inclusion Criteria:

* All subjects between the ages of 18 and 70 with chronic hepatitis B and under the oral anti-virus treatment followed at the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, China, will be offered entry into this study. The diagnosis of chronic Hepatitis B will be based on that they had been positive for hepatitis B surface antigen (HBsAg) for at least six months, and were positive for HBeAg or negative for HBeAg with detectable HBV DNA at screening.
* No evidence of HCC on entry imaging study.
* Model for End Stage Liver Disease (MELD) score under 22 (a MELD score over 22 would predict a 3 month mortality rate of approximately 20%).
* Not currently participating in another intervention study.
* Not pregnant or lactating, and willing to use effective contraception during study period.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Ability to provide written informed consent according to national/local regulations.

Exclusion Criteria:

* evidence of hepatocellular carcinoma within 6 months after enrollment,
* a serum alanine aminotransferase level more than 10 times the upper limit of normal,
* an elevated serum creatinine level,
* any diagnosis of kidney stones,
* a diagnosis of hyperparathyroidism or other serious disturbance of calcium metabolism in the past 5 years,
* any evidence of autoimmune hepatitis, coinfection with hepatitis C or D virus or human immunodeficiency virus,
* other serious concurrent illness (e.g., alcoholism, uncontrolled diabetes, or cancer),
* treatment with immunomodulatory within the 6 months before screening,
* treatment with any investigational drug within the 30 days before the study began.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum levels of 25-hydroxy vitamin D | at baseline, and at 6 and 12 months
  Change in serum levels of 25-hydroxyvitamin D at 6 months and 12 months compared to baseline

SECONDARY OUTCOMES:
Change in serum creatinine | at baseline, and at 6 and 12 months
  Change in serum creatinine at 6 months and at 12 months compared to baseline
Change in fibrosis score | at baseline, and at 6 and 12 months
  Change in fibrosis score at 6 months and at 12 months compared to baseline. The investigators use Fibroscan to get the score of fibrosis.
Number of participants on Vitamin D treatment with adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yutian Chong, MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Result] Dalhoff K, Dancey J, Astrup L, Skovsgaard T, Hamberg KJ, Lofts FJ, Rosmorduc O, Erlinger S, Bach Hansen J, Steward WP, Skov T, Burcharth F, Evans TR. A phase II study of the vitamin D analogue Seocalcitol in patients with inoperable hepatocellular carcinoma. Br J Cancer. 2003 Jul 21;89(2):252-7. doi: 10.1038/sj.bjc.6601104. PMID 12865912
- [Result] Ding EL, Mehta S, Fawzi WW, Giovannucci EL. Interaction of estrogen therapy with calcium and vitamin D supplementation on colorectal cancer risk: reanalysis of Women's Health Initiative randomized trial. Int J Cancer. 2008 Apr 15;122(8):1690-4. doi: 10.1002/ijc.23311. PMID 18092326
- [Result] Krishnan AV, Feldman D. Mechanisms of the anti-cancer and anti-inflammatory actions of vitamin D. Annu Rev Pharmacol Toxicol. 2011;51:311-36. doi: 10.1146/annurev-pharmtox-010510-100611. PMID 20936945
- [Result] Woo TC, Choo R, Jamieson M, Chander S, Vieth R. Pilot study: potential role of vitamin D (Cholecalciferol) in patients with PSA relapse after definitive therapy. Nutr Cancer. 2005;51(1):32-6. doi: 10.1207/s15327914nc5101_5. PMID 15749627
- [Result] Amir E, Simmons CE, Freedman OC, Dranitsaris G, Cole DE, Vieth R, Ooi WS, Clemons M. A phase 2 trial exploring the effects of high-dose (10,000 IU/day) vitamin D(3) in breast cancer patients with bone metastases. Cancer. 2010 Jan 15;116(2):284-91. doi: 10.1002/cncr.24749. PMID 19918922
- [Result] Sherman MH, Yu RT, Engle DD, Ding N, Atkins AR, Tiriac H, Collisson EA, Connor F, Van Dyke T, Kozlov S, Martin P, Tseng TW, Dawson DW, Donahue TR, Masamune A, Shimosegawa T, Apte MV, Wilson JS, Ng B, Lau SL, Gunton JE, Wahl GM, Hunter T, Drebin JA, O'Dwyer PJ, Liddle C, Tuveson DA, Downes M, Evans RM. Vitamin D receptor-mediated stromal reprogramming suppresses pancreatitis and enhances pancreatic cancer therapy. Cell. 2014 Sep 25;159(1):80-93. doi: 10.1016/j.cell.2014.08.007. PMID 25259922